CLINICAL TRIAL: NCT00000897
Title: The Effect of Oral and Injectable Contraceptives (Norethindrone/Ethinyl Estradiol, Medroxyprogesterone Acetate) and Gender on Plasma and Intracellular Zidovudine Pharmacokinetics
Brief Title: A Study to Evaluate the Effects of Different Methods of Birth Control on the Drug Actions of Zidovudine (an Anti-HIV Drug) in HIV-Positive Women and to Compare Zidovudine Metabolism in Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: ACTG 317; AACTG 317
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-03

CONDITIONS: HIV Infections
Keywords: Drug Interactions; Zidovudine; Sex Factors; Reverse Transcriptase Inhibitors; Contraceptives, Oral; Progestational Hormones, Synthetic; Anti-HIV Agents; Viral Load; Estrogens
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
The purpose of this study is to look at the effects of different methods of birth control (oral and injectable) on how the body absorbs, makes available, and removes zidovudine (ZDV). This study will also evaluate the differences in men and women in how the body absorbs, makes available, and removes ZDV.

Past research has shown that the effectiveness of ZDV as an anti-HIV drug might be decreased in individuals who use certain methods of birth control. ZDV may also have different effects in men compared to women.

DETAILED DESCRIPTION:
Oral contraceptives have been shown to substantially enhance the glucuronidation of several compounds. One study reported enhanced glucuronidation of oxazepam, a compound that is conjugated via the same UDP-glucuronyl transferase isozyme responsible for ADV glucuronidation, suggesting that ZDV metabolism may be altered by concomitant oral contraceptive use. This potential enhancement of ZDV metabolism by oral contraceptives is expected to result in decreased plasma levels of the parent compound which may lead to diminished clinical efficacy in women using these drugs. It remains unclear whether the progesterone and/or estrogen component of oral contraceptives results in the observed glucuronidation changes.

This open-label, pharmacokinetic trial is conducted in 2 steps. [AS PER AMENDMENT 6/12/01: The Depo-Provera IM group in Step 2 is filled. Female patients who choose to participate in Step 2 may enroll only in the Ortho-Novum 1/35 PO group.] [AS PER AMENDMENT 11/13/00: Female patients may choose to participate in Step 1 alone or both Steps 1 and 2.] Male patients may participate in Step 1 only as the control arm of the study. In Step 1, patients are stratified by sex; in Step 2, female patients are stratified by their choice of contraception (i.e., oral norethindrone/ethinyl estradiol [Ortho-Novum 1/35] or injectable medroxyprogesterone acetate [Depo-Provera]).

Step 1 (males and females): At entry, all patients are randomized to receive ZDV either orally or orally and intravenously (IV) on Days 7 and 8. Female patients begin the study (Day 0) between days 10-18 after the first day of their last menstrual period (LMP) (Cycle 1). At time of enrollment, female patients [AS PER AMENDMENT 11/13/00: who plan to participate in Step 2] choose the form of birth control instituted in Step 2: Depo-Provera or Ortho-Novum 1/35. Male patients may enter Step 1 at any time. Patients continue taking their other pre-study antiretroviral drugs during Step 1. [AS PER AMENDMENT 6/3/99: Patients taking nelfinavir may participate only in the Depo-Provera arm.] Days 0-6: All patients receive oral ZDV. Day 7: Patients are randomized to receive:

Arm 1 (females): oral ZDV for a total of 3 doses. Arm 2 (females): ZDV IV, then ZDV orally for a total of 2 oral doses. Arm 3 (males): control arm. Half of the male patients receive ZDV as in Arm 1 and the other male patients receive ZDV as in Arm 2.

Day 8: Patients on all 3 arms receive the alternate form of ZDV to that received on Day 7. Day 9: Female patients resume their pre-study method of administration of ZDV. Male patients conclude their participation in the study on Day 8.

Step 2 (females [AS PER AMENDMENT 11/13/00: opting to participate in Step 2]): At the onset of their second menstrual period (Cycle 2) since starting study, female patients start their choice of Ortho-Novum 1/35 or intramuscularly administered Depo-Provera [AS PER AMENDMENT 6/12/01: Enrollment for Depo-Provera is closed]. Contraceptive therapy continues throughout Step 2. Step 2 Days 0-6: Between days 7-11 [AS PER AMENDMENT 6/3/99: Between days 7-18] of the third menstrual cycle (Cycle 3) since starting study, female patients continue their pre-study antiretroviral therapy (as done in Step 1) and begin another course of ZDV standard therapy 3 times daily. Days 7-8: Patients receive the original method of administration of ZDV (as randomized at study entry). Female patients return for a final safety visit within 1 week of completing study Day 8 of Step 2.

ELIGIBILITY:
Inclusion Criteria

Men and women may be eligible for this study if they:

* Are HIV positive.

Women may be eligible for this study if they:

* Have regular periods and a normal gynecological exam, (including a Pap smear and mammogram).
* Enter the study between Days 10 and 18 of the first day of their last period.
* Are willing to use either the Pill or Depo-Provera as birth control.
* Have a negative pregnancy test within 14 days prior to study.

Exclusion Criteria

Men and women will not be eligible for this study if they:

* Cannot take ZDV for any reason.
* Have cancer.
* Are taking stavudine.

Women will not be eligible for this study if they:

* Cannot take the Pill or Depo-Provera.
* Are pregnant or nursing.
* Are receiving nelfinavir and want to enroll in Step 2.
* Have a history of chronic high blood pressure, thrombophlebitis, and/or pulmonary emboli if participating in Step 2 of the study.

(This study has been changed so that women with certain criteria are excluded from participating in Step 2.)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42
Dates: Primary Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Aweeka, Study Chair
Locations (6):
- United States (6):
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Univ of Washington, Seattle, Washington